CLINICAL TRIAL: NCT02063022
Title: Phase III Study on Efficacy of Dose Intensification in Patients With Non-metastatic Ewing Sarcoma.
Brief Title: Efficacy of Dose Intensification in Patients With Non-metastatic Ewing Sarcoma
Acronym: EW-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Italian Sarcoma Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISG/AIEOP EW-1
Record Dates: First submitted 2013-02-21; First posted 2014-02-14 (Estimated); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Ewing's Sarcoma
Keywords: Non metastatic Ewing's Sarcoma
MeSH Terms: conditions — Sarcoma, Ewing | interventions — Vincristine; Dactinomycin; Doxorubicin; Ifosfamide; Cyclophosphamide; Etoposide; Busulfan; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard treatment (as per ISG SSG III protocol) (Active Comparator): Standard treatment for non metastatic Ewing's Sarcoma (as defined by the ISG/SSG III protocol).
  It is based on a 6 drugs pre-local treatment (Vincristin, dactinomycin, cyclophosphamide,ifosfamide,etoposide and doxorubicin) followed by local treatment (surgery and/or radiotherapy)and by a maintenance treatment based on induction response
  Interventions: Drug: Standard treatment (as per protocol ISG SSG III)
- Intensified treatment (Experimental): Dose intense treatment for non metastatic Ewing's Sarcoma It is based on a 3 drug pre-local treatment (Vincristin, ifosfamide and doxorubicin)followed by local treatment (surgery and/or radiotherapy)and by a maintenance treatment based on induction response
  Interventions: Drug: Intensified chemotherapy

INTERVENTIONS:
Drug: Standard treatment (as per protocol ISG SSG III) — Induction treatment with: 4 cycle of Vincristine (9mg/,2), Dactinomycin (6mg/m2), Doxorubicin (160mg/m2), Cyclophosphamide (2.4g/m2), Ifosfamide (18g/M2) and Etoposide (450mg/m2) given every 3 weeks Maintenance treatment for poor responder (25 weeks): Vincristine (12mg/m2), Dactinomycin (1.5mg/m2), Doxorubicin (320mg/m2), Ifosfamide (27g/m2), Cyclophosphamide (8.8g/m2), Etoposide (1.5g/m2) and peripheral Cells Steam Transplant after Busulfan and Melphalan treatment Maintenance treatment (37 week) for good responder: Vincristine (18mg/m2), Dactinomycin (6mg/m2), Doxorubicin (400mg/m2), Ifosfamide (72g/m2), Cyclosphosphamide(6g/m2), Etoposide (1.8 g/m2)
  Other Names: Vincristine; Dactinomycin; Doxorubicin; Ifosfamide; Cyclophosphamide; Etoposide; Busulfan; Melphalan
  Arms: Standard treatment (as per ISG SSG III protocol)
Drug: Intensified chemotherapy — * Induction treatment with: 4 cycle of Vincristine (10.5 mg/m2), Doxorubicin (320 mg/m2) and Ifosfamide (36 mg/m2) given every 3 weeks
  * Maintenance treatment for poor responder (25 weeks): Vincristine (12mg/m2), Doxorubicin (400mg/m2), Ifosfamide (63g/m2), Cyclophosphamide (4g/m2), Etoposide (1.5g/m2) and Cells Steam Transplant after Busulfan and Melphalan treatment
  * Maintenance treatment (25 week) for good responder: Vincristine (12mg/m2), Doxorubicin (400mg/m2), Ifosfamide (72g/m2), Etoposide (1.8g/m2)
  Other Names: Vincristine,; Doxorubicin; Ifosfamide; Cyclophosphamide; Etoposide; Busulfan; Melphalan
  Arms: Intensified treatment

SUMMARY:
Controlled, randomized phase III study, with the intent of optimizing the treatment of not metastatic Ewing Sarcoma. The patients will be randomized into 2 arms: standard treatment vs intensive treatment. Both arms will receive an induction treatment followed by surgery (wherever is possible) and/or radiotherapy. The maintenance treatment will be different on the basis of the response to the induction treatment (good or poor)

DETAILED DESCRIPTION:
Eligible patients with non metastatic Ewing's Sarcoma will be randomized into 2 different arms: standard treatment arm A (based on the ISG/SSG III protocol) or into the experimental arm B(chemotherapy with dose intensification and shorter length of treatment).

Both arm will receive an induction treatment with higher dose intensity of doxorubicin and ifosfamide in Arm B.

After the induction treatment all the patient will undergo to local treatment (surgery and/or radiotherapy)that will be followed by a maintenance therapy.

The maintenance therapy will be different for both arms and, within each arm, on the basis of the response (histologically evaluated) of the pre-local treatment therapy.

Maintenance for Arm A: Poor responders will undergo to stem cells apheresis and their reinfusion after treatment with high doses of Busulfan and Melphalan 25 weeks.

Good responders will receive a 6 drugs maintenance treatment for 37 weeks (as per standard ISG/SSG III protocol)

Maintenance for Arm B: Poor responders will undergo to stem cells apheresis and their reinfusion after an intensified treatment with high doses of Busulfan and Melphalan (25 weeks).

Good responders will receive a maintenance treatment for 25 weeks

The primary aim of the study is to assess the Event Free Survival (EFS) that is expected to be similar in both arms

The secondary objectives are:

To assess if the induction treatment in Arm B is able to increase the percentage of good responders compared to those who receive standard treatment.

To assess the toxicity and the Quality of Life related to the chemotherapy treatment

ELIGIBILITY:
Inclusion Criteria

* Ewing Sarcoma or PNET diagnosis centrally confirmed
* Age ≤ 40 years
* Absence of evident metastasis or lung met < 0.5 cm Presence of skip metastasis in the bone compartment of the primary tumor is to be considered as local disease and not metastatic.
* Adeguate bone marrow, hepatic and renal function
* Left Ventricular Ejection Fraction > 50%
* No primary Ewing Sarcoma treatments (both chemotherapy and/or radiotherapy)
* Voluntarily signed an informed consent form
* Radiological and histological documentation available for central review.

Exclusion Criteria

* Presence of lung or extra-pulmonary lesions
* Bone Marrow involvement
* In case of chest disease: presence of plural effusion
* Elapsed time between histological diagnosis and chemotherapy start, more than 4 weeks
* Any medical contraindication to the use of the study drugs
* Any psychological or social conditions that can compromise the protocol compliance and/or follow-up
* Previous malignancies (excluded in situ cervix carcinoma)

Max Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 278 (Actual)
Dates: Start 2009-01-22 (Actual); Primary Completion 2022-04-14 (Actual); Study Completion 2022-04-14 (Actual)

PRIMARY OUTCOMES:
Event Free Survival (EFS) | 5 years
  The EFS (event defined as Progressive Disease , onset of local relapse and/or metastasis, death due to chemotherapy toxicity or for other causes) will be calculated from the first treatment day up to the event onset or to last follow-up

SECONDARY OUTCOMES:
Disease Free Survival (DFS) | expected average 3 years
  The DFS will be calculated from the day that the patient will be free from disease (surgery date and/or radiotherapy completion) up to the date of progression disease or last follow-up
Metastasis Free Survival | expected average 2 years
  The Metastasis free Survival will be evaluated from the time of disease free (surgery performed and/or radiotherapy completed) to the onset of distance metastasis or last follow-up
Overall Survival (OS) | expected average 5 years
  The OS will be evaluated for the start treatment day to the day of death (for any causes)

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Luksch, MD, Principal Investigator — Italian Sarcoma Group
Locations (14):
- Italy (14):
  - Centro di Riferimento Oncologico - Unit of Medical Oncology, Aviano, Pordenone
  - I.R.C.C. - Unit of Medical Oncology, Candiolo, Torino
  - IRCCS materno infantile Burlo Garofolo, Trieste, T
  - Azienda Ospedaliero Universitaria Consorziale Policlinico - Bari, Bari
  - Istituto Ortopedico Rizzoli, Bologna
  - A.O. Universitaria Meyer, Florence
  - Istituto Giannina Gaslini, Genova
  - FONDAZIONE IRCCS Istituto Nazionale dei Tumori, Milan
  - Azienda Ospedaliera Universitaria "Federico Ii" ., Napoli
  - Azienda Ospedaliera di Padova, Padua
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Istituto Nazionale Tumori Regina Elena - Unit of Medical Oncology I, Roma
  - Ospedale Pediatrico Bambin Gesu', Roma
  - Ospedale Infantile Regina Margherita - Unit of Paediatric Oncoematology, Torino

REFERENCES:
- [Background] S. Ferrari, T. Alvegard, R. Luksch, A. Tienghi, K. S. Hall, G. Bernini, A. Brach del Prever, P. Picci, G. Bacci, S. Smeland Non-metastatic Ewing's family tumors: High-dose chemotherapy with stem cell rescue in poor responder patients. Preliminary results of the Italian/Scandinavian ISG/SSG III protocol. J Clini Oncol, 2007 ASCO Annual Meeting Proceedings Vol 25 (June 20 Suppl), 2007: 10014
- [Derived] Luksch R, Palmerini E, Milano GM, Paioli A, Asaftei S, Barretta F, Puma N, Cesari M, Tirtei E, Podda M, Pierobon M, Manzitti C, Ferraresi V, Tamburini A, Bertulli R, Di Pinto D, Mascarin M, Grignani G, Coccoli L, Rabusin M, De Leonardis F, Gambarotti M, Parafioriti A, Cammelli S, Vennarini S, Ferrari S, Donati DM, Bastoni S, Massimino M, Fagioli F, Ibrahim T. Intensified Induction Therapy for Newly Diagnosed, Localized Skeletal Ewing Sarcoma (ISG/AIEOP EW-1): A Randomized, Open-Label, Phase 3, Non-Inferiority Trial. Pediatr Blood Cancer. 2025 Apr;72(4):e31551. doi: 10.1002/pbc.31551. Epub 2025 Jan 20. PMID 39833645